CLINICAL TRIAL: NCT03055078
Title: Evaluation of Safety and Efficacy in Patients With Aplastic Anemia by Transplantation of Umbilical Cord Derived Mesenchymal Stem Cells
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Aplastic Anemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17277787D-AA
Record Dates: First submitted 2017-02-04; First posted 2017-02-16 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mesenchymal stem cells (Experimental): According to the inclusion and exclusion criteria, selected patients were divided into a cell therapy group and a control group. Umbilical cord derived mesenchymal stem cells at a dose of 100-300 million by intravenous infusion.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Patients in the cell treated group were given umbilical cord derived mesenchymal stem cells by intravenous infusion besides conventional therapy. There was only conventional treatment in the control group. All patients after treatment for 1months, 3months, 6months and 9months were evaluated respectively the therapeutic effect.

SUMMARY:
This study is to evaluate the safety and efficacy of Umbilical Cord Derived Mesenchymal Stem Cells transplantation in aplastic anemia.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is a disorder thought to be caused by an immune-mediated bone marrow failure. Not all people with AA are eligible for today's standard treatments. One new treatment approach uses umbilical cord derived mesenchymal stem cells-specialized cells capable of developing into other types of cells-to provide the basis for clinical application. The aim of the present study is to investigate the safety and efficacy of vein infusion of allogeneic mesenchymal stem cells in patients with AA .

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AA according to established criteria in 2010
2. Age from 14 to 60 years
3. Suffering from AA within six months
4. No serious infection or acute hemorrhage.
5. Left ventricular ejection fraction (LVEF) ≥ 50%
6. No acute infectious diseases.
7. Understanding and willingness to sign a written informed consent document.
8. Eastern Cooperative Oncology Group(ECOG) score of 0-2pionts.

Exclusion Criteria:

- Patients with AA have to be disqualified from this study if any of the following is applicable.

1. Severe aplastic anemia(SAA) with severe infection.
2. Severe aplastic anemia(SAA) with active hemorrhage.
3. Severe heart attack, liver and kidney disease following serious complications
4. Patients with allergic constitution.
5. Pregnancy and lactation.
6. Accompanied by malignant tumors and other clonal disease.
7. Patients with active tuberculosis, acute sever hepatitis or infectious period of diseases.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin levels in peripheral blood | Post cell transplantation: 9months
  The recovery of bone marrow erythrocyte is evaluated by hemoglobin levels (g/L) in peripheral blood.

SECONDARY OUTCOMES:
The number of red blood cell in peripheral blood | Post cell transplantation: 1, 3, 6, 9months
  The improvement of bone marrow erythrocyte is evaluated by red blood cell count (×10^12/L) in peripheral blood.
The number of granulocyte in peripheral blood | Post cell transplantation: 1, 3, 6, 9months
  The recovery of bone marrow granulocyte is evaluated by granulocyte count (×10^9/L) in peripheral blood.
The number of white blood cell in peripheral blood | Post cell transplantation: 1, 3, 6, 9months
  The improvement of bone marrow granulocyte is evaluated by white blood cell count (×10^9/L) in peripheral blood.
The evaluation of bone marrow megakaryocytic series | Post cell transplantation: 1, 3, 6, 9months
  The status of megakaryocytic series is evaluated by platelet count (×10^9/L) in peripheral blood.
adverse reaction | Post cell transplantation: 1, 3, 6, 9months
  Adverse reaction includes temperature changes(℃), the change of blood pressure(mmHg) and allergic reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — The First Hospital of Hebei Medical University; Qingchi Liu, Doctor, Study Director — The First Hospital of Hebei Medical University; Quanhai Li, Doctor, Study Director — The First Hospital of Hebei Medical University; Xiaohui Jia, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Xianyun Wang, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Fan Zhang, Bachelor, Principal Investigator — The First Hospital of Hebei Medical University; Yang Shen, Master, Principal Investigator — The First Hospital of Hebei Medical University; Bing Ma, Master, Principal Investigator — The First Hospital of Hebei Medical University; Wanyi Yin, Master, Principal Investigator — The First Hospital of Hebei Medical University; Dan Zhao, Master, Principal Investigator — The First Hospital of Hebei Medical University; Bojian Sun, Master, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No